CLINICAL TRIAL: NCT00288977
Title: Islet Transplantation in Type 1 Diabetic Recipients of Renal Allografts, Using the Edmonton Protocol
Brief Title: Islet Transplantation in Type 1 Diabetic Recipients of Kidney Transplants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Martha Pavlakis, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001P001702
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Kidney Transplantation
Keywords: Diabetes; Islet Transplantation
MeSH Terms: conditions — Diabetes Mellitus

ARMS (1):
- islet cell transplant (Experimental)
  Interventions: Procedure: Islet Infusion

INTERVENTIONS:
Procedure: Islet Infusion

SUMMARY:
Study hypothesis is that we can reproduce results of islet transplantation in type one diabetics in patients with a kidney transplant.

DETAILED DESCRIPTION:
This trial is designed to replicate the protocol currently being tested by the Immune Tolerance Network (ITN) in a population of patients that have been previously transplanted (recipients of functioning renal allografts) and are therefore immunosuppressed.

The data will be generated using substantially identical techniques for islet preparation, re transplantation with additional islets to meet the minimum islet cell mass, and an identical steroid-free post-transplant regimen utilizing sirolimus, low dose tacrolimus, and daclizumab.

3.1. Primary and secondary endpoints and additional measures

Study efficacy endpoints and additional measures are described in the following subsections. Measures relating to the islet preparation quality (Section 3.1.3) and other variables relating to key cellular and genetic markers (Section 3.1.4) followed during the study are not considered clinical outcome variables. Details describing requirements for efficacy testing are found in Section 6.1. Safety measures are described in Section 7.

3.1.1. Primary endpoint

The primary endpoint for this study is independence from insulin injections with adequate control of blood glucose in subjects with Type 1 diabetes at one year post final transplant. Subjects will be considered as a success when at the one year assessment they are not using insulin, they have a HbA1c <6.5% and they achieve fasting glucose levels not exceeding 7.8 mmol/L (140 mg/dL) more than three times in a week (using the morning fasting glucose level), and not exceeding two hour post-prandial (using any post meal glucose level) values of 10 mmol/L (180 mg/dL) more than four times in a week. A subject will still be considered a success if an intercurrent illness or other event (e.g., high tacrolimus level) causes a participant to require insulin use for a period not exceeding a total of 14 days, and assessment after this event demonstrates insulin independence and adequate glucose control as defined above. This assessment must be completed no later than two weeks after the scheduled one year assessment.

3.1.2. Secondary parameters

Secondary parameters that support the primary goal of the investigation will be assessed at generally the same intervals as the primary endpoint, with some taken more or less frequently as indicated in detail in Sections 5.2 and 6.1. Additional clinical measurements are also taken during the study that are not considered endpoints for formal analyses, but are to be carefully followed as a part of the study. The schedule for these additional elements is listed in Sections 5.2, 6.2 and 7.2. The secondary variables include the following measures:

1. Basal C-peptide levels
2. HbA1C levels
3. Glucose tolerance
4. C-peptide response to arginine
5. MAGE improvement
6. Mixed Meal Test
7. Durability of insulin independence and adequate blood glucose control

3.1.3. Islet quality endpoints

Islet cell preparations for each transplant will be assessed using the following elements:

1. Islet yield per isolation used for clinical transplantation, expressed as i) total islet equivalents and ii) islet equivalents per kg recipient body weight.
2. Islet viability, as assessed by a fluorescent dye inclusion/exclusion assay to assess metabolic activity and membrane integrity.
3. In vitro islet responsiveness to glucose challenge, as measured by 2-hour static incubation following 12-24 hour culture at 37º C in CMRL 1066 (10% FCS, 25 mmol HEPES). A stimulation index, a ratio of insulin secretion during high glucose over insulin secretion during low basal secretion is calculated as an index of islet function.
4. Islet cell immunohistochemical composition and purity assessment, (as determined by JDRF Center for Islet Transplantation at Harvard Medical School - Islet Morphology Core Laboratory)
5. Evidence of no microbial contamination, as documented by a negative Gram stain of the islet preparation immediately pre-transplant, and by negative microbial cultures reported after at least 5 days incubation for aerobes, anaerobes, fungi.
6. Evidence of a low endotoxin content of the final islet preparation.

3.1.4. Cellular and genetic markers

Samples will be collected before and after transplant for immunologic studies to be processed in the laboratories of Dr. Terry Strom at the Beth Israel Deaconess Medical Center and Dr. Mohamed Sayegh at the Brigham and Women's Hospital.

These include:

1. Alteration in autoimmune markers for GAD65, ICA512, and mIAA, comparing blood samples drawn pre-transplant and 3, 6, 9, 12, 24 and 36 months after final transplant.
2. Changes in autoantibody and other immune markers comparing blood samples drawn pre-transplant and 3, 6, 12, 24, and 36 months after final transplant
3. Samples will also be taken for future laboratory and genetic studies comparing blood samples drawn pre-transplant and usually 3, 6, and 12 months after final transplant.

3.2. Description of trial design and schematic diagram of procedures and stages

Because this is an open-label, single-arm study, a schematic diagram of the design is omitted for simplicity. For a general description of the trial design, please refer to Section 2. A tabular listing of visit schedules and tests is found in Appendix 1.

3.3. Measures to minimize bias

This study is an open-label feasibility study with definitive clinical endpoints of insulin independence, blood glucose and C peptide production as measures of procedural success. As donor islets become available the appropriate ABO compatible blood types will be matched to eligible participants. Clinical investigators are not masked to treatment assignment or follow up assessment information for this pilot study.

3.4. Description of trial treatments and dosage regimen & labeling

Each islet cell transplantation procedure under this protocol is derived from an individual donor pancreas, processed for immediate transplantation. All containers and components are appropriately labeled during preparation. Each final islet preparation released for use is labeled to indicate its identity and date of preparation. Records regarding donor identity will be kept in a coded manner for quality control purposes and will be kept absolutely confidential in accordance with standard procedures.

3.4.1. Islet Infusion(s)

A target total of > 10,000 IE/kg recipient body weight will be infused via a percutaneous transhepatic catheter inserted into the portal vein (see Section 1.4.2). This will in all likelihood require more than one islet infusion to achieve this goal. The first infusion must contain at least 5,000 IE/kg recipient body weight. In the event that a subject does not achieve insulin-independence with normoglycemia after two fresh islet infusions, a third transplant may be considered as described in Section 5.1.

3.4.2. Immunosuppressive Therapy

Beginning with the initial transplant, a immunosuppressive regimen will be administered to all subjects. Subjects will receive initial doses of daclizumab, sirolimus, and low dose tacrolimus according to the following schedule.

3.4.2.1. Daclizumab regimen

Daclizumab will be administered at a dose of 1 mg/kg peripheral IV given immediately pre-transplant, and at 2, 4, 6, and 8 weeks after transplant, for a total of 5 doses (over 8 weeks). If a subsequent islet infusion is required beyond this induction period, then a further 5 dose course of daclizumab will be given according to the same schedule. If the second (or third) transplant occurs and no daclizumab was given in the preceding 7 days, then the dosing regimen will begin at the time of transplant. If daclizumab has been administered within the past 7 days, then the dose at transplant is omitted, and the first dose given 2 weeks post transplant.

3.4.2.2. Sirolimus regimen

All patients enrolled in this trial will already be on Sirolimus therapy. If needed, the dose will be increased to 0.1 mg/kg/day PO and adjusted to the target range of 12-15 ng/ml for the 3 months following the most recent islet infusion. After three months following last transplant, the target whole blood level will be lowered to 7-10ng/mL.

3.4.2.3. Tacrolimus regimen

All patients enrolled in this trial will already be on Tacrolimus therapy. As soon as trough levels are available, the dose will be adjusted to the target range of 3-6 ng/ml throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Enrolling subjects must have Type 1 diabetes mellitus for more than 5 years, complicated by renal failure requiring a kidney transplant. The complicating situations are:

1. Reduced awareness of hypoglycemia,
2. Metabolic lability/instability,
3. Despite efforts at optimal glucose control, progressive secondary complications of diabetes as defined by:

i) Retinopathy- ii) Nephropathy- or

iii) Neuropathy-

Exclusion Criteria:

1. Severe co-existing cardiac disease, characterized by any one of these conditions:

   * recent myocardial infarction (within past 6 months), or
   * angiographic evidence of non-correctable coronary artery disease, or
   * evidence of ischemia on functional cardiac exam (•
2. Active alcohol or substance abuse-includes cigarette smoking (

   * Failure to fulfill major work, school, or home responsibilities;
   * Drinking in situations that are physically dangerous, such as while driving a car or operating machinery;
   * Recurring alcohol-related legal problems, such as being arrested for driving under the influence of alcohol or for physically hurting someone while drunk;
   * Continued drinking despite having ongoing relationship problems that are caused or worsened by the effects of alcohol.
3. Psychiatric disorder making the subject not a suitable candidate for transplantation,
4. History of non-adherence to prescribed regimens
5. Active infection including hepatitis C, hepatitis B, HIV, or TB (or under treatment for suspected TB)
6. Any history of malignancy except squamous or basal skin cancer
7. BMI > 26 kg/m2 or body weight > 70 kg for females and > 75kg for males at the screening visit. (An allowance for weight gain of up to +2 kg body weight is permitted between the screening visit and actual transplant. No transplant can be given to a female subject weighing > 72 kg or a male subject weighing > 77kg on the day of transplant. See Section 5.1 for minimum islet equivalent infusion requirements per recipient body weight.)
8. C-peptide response to arginine stimulation (5 gm I.V.) (any C-peptide ≥ 0.3 ng/mL at 2, 3, 4, 5, 7 and 10 min post infusion)
9. Inability to provide informed consent
10. Age less than 18 or greater than 65 years
11. Serum creatinine > 1.8 mg/dL, In addition, there must be no change in serum creatinine of > 0.4 mg/dl in the last 6 months.
12. Baseline Hb < 10.5 gm/dL in women, or < 13 gm/dL in men
13. Baseline LFT's outside of normal range with the exception of Gilberts Syndrome. n. Presence of gallstones (subjects may be eligible two weeks after a laparoscopic cholecystectomy ).

o. Hemangioma in liver on baseline ultrasound exam

p. Untreated proliferative retinopathy

q. Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast feeding

r. Evidence of sensitization as determined by a general PRA with reactivity > 20%. t. Insulin requirement > 0.7 IU/kg/day

s. HbA1C > 12%

t. Inability to complete all scheduled visits during screening and post-transplant follow-up

u. Hyperlipidemia (fasting LDL cholesterol > 130 mg/dL, treated or untreated; and/or fasting triglycerides > 200 mg/dL).

v. Under treatment for a medical condition requiring chronic use of steroids at a dose > prednisone 5 mg/day w. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT INR > 1.5 x. Addison's disease.y. EBV- negative subjects (use EBNA test for screening) to reduce potential risk of EBV infection for previously unexposed recipient.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2000-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
independence from insulin injections with adequate control of blood glucose in subjects with Type 1 diabetes at one year post final transplant | one year post final islet cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Martha Pavlakis, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Joslin Diabetes Clinic

IPD SHARING:
Plan to Share IPD: No